CLINICAL TRIAL: NCT04892394
Title: Determining the Effect of Video Information on the Dental Anxiety Levels of the Endodontic Patients: A Randomized Clinical Trial
Brief Title: Effect of Video Information on the Dental Anxiety Levels of the Endodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Hicran Dönmez Özkan, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ADÜDHF 2019/071
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Dental Anxiety
Keywords: Video information; Electrodermal activity; Endodontic treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Detailed visual video information was given to the video group patients before endodontic treatment by the clinician.
  Interventions: Other: Information Types Before Endodontic Treatment
- Control Group (Experimental): Basic verbal information was given to the control group patients before endodontic treatment by the clinician.
  Interventions: Other: Information Types Before Endodontic Treatment

INTERVENTIONS:
Other: Information Types Before Endodontic Treatment — The first aim of this study is to compare the effect of detailed video information or basic verbal information on the anxiety levels of patients by using anxiety scales before treatment. The second aim is to evaluate the effect of pretreatment video or verbal information on the stress level occurring in patients during the endodontic treatment steps by using electrodermal activity. The third aim is to investigate the relationship between patients' pretreatment anxiety levels and socio-demographic characteristics which are thought to play a role in anxiety's etiology.

SUMMARY:
This study compared the effect of the detailed video visual information and basic verbal information on patients' anxiety levels (using anxiety scales) before endodontic treatment and stress levels (using electrodermal activity method) during endodontic treatment.

DETAILED DESCRIPTION:
Patients (n=120) aged between 18-65 with single-rooted teeth with the single canal that diagnosed with asymptomatic irreversible pulpitis and/or pre-prosthetic root canal treatment were included in this study. Patients were randomly divided into two groups after completing anxiety scales and socio-demographic/dental habits form. Before the treatment, visual video information was given to the video group patients, while the control group patients were routinely informed verbally. The stress levels during the endodontic treatment process were recorded by placing a electrodermal activity measurement device on the wrists of the patients. Anxiety scales and feedback-satisfaction forms were administered to all patients after the treatment process.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 - 65 years of ages
2. Patients with healthy (ASA 1) and mild systemic disease (ASA 2) according to ASA classification
3. Patients with no mental disorders in their medical history
4. Patients who do not have a psychiatric disorder that they have started, and who do not use psychotherapeutic drugs.
5. Literate and not visually impaired patients
6. Patients presenting with single-rooted teeth with a single root canal diagnosed with asymptomatic irreversible pulpitis or single-rooted vital teeth with a single root canal requiring root canal treatment due to prosthetic reasons

Exclusion Criteria:

1. Patients who refuse to participate this study
2. Patients have existing pain caused by another tooth
3. Patients with dermatological disease in the medical histories
4. Medically compromised patients (with immunosuppressive/systemic diseases, patients on medications)
5. The presence of spontaneous pain, swelling, or fistula in the relevant tooth
6. Teeth whose working length cannot be reached due to calcification and step formation in the root canal
7. The presence of foreign material in the root canal that prevents entry (broken instrument, post)
8. The presence of advanced periodontal disease (probing depth > 4 mm) or root fracture in the relevant tooth
9. Patients using pain medication on the same day before treatment (within 24 hours)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
Anxiety level comparison after endodontic treatment with two preoperative information types | Immediately after treatment
  Modified Dental Anxiety Scale (MDAS) was used to assess anxiety levels. The Modified Dental Anxiety Scale (MDAS) consisted of 5 questions ranging from 5 (no anxiety) to 25 (highest anxiety level). Every patient was asked to mark his or her perceived dental anxiety level on the line.
Anxiety level comparison after endodontic treatment with two preoperative information types | Immediately after treatment
  State Anxiety Scale (STAI-S) was used to assess anxiety levels. The STAI scales consisted of two scales, each with 20 questions, with a total score between 20 and 80. Every patient was asked to mark his or her perceived dental anxiety level on the line.
Anxiety level comparison after endodontic treatment with two preoperative information types | Immediately after treatment
  The Visual Analogue Scale (VAS) was a scale consisting of a horizontal straight line 0-100 mm long with words describing the two extremes of the condition to be measured at both ends (i.e. zero - no anxiety, maximum - most severe anxiety). Every patient was asked to mark his or her perceived dental anxiety level on the line.
Electrodermal activity level comparison during endodontic treatment with two preoperative information types | During endodontic treatment process
  At the beginning of the endodontic treatment, the GSR device was attached to the patient's preferred wrist, and the measuring tapes of the device were placed on the patient's proximal phalanges of the index and middle finger. One-visit endodontic treatment was divided into 7 steps (anesthesia, cavity preparation, rubber dam placement, determination of root canal length, root canal shaping, root canal filling, coronal restoration and finishing) and recorded. All data transmitted to the computer via a wireless connection by a software program were recorded at the end of the treatment.

SECONDARY OUTCOMES:
Evaluation of the relationship between patients' pretreatment anxiety levels and socio-demographic characteristics and dental treatment habits | Before Endodontic Treatment
  The patients were asked to fill in anxiety scales and sociodemographic/dental habits forms. Modified Dental Anxiety Scale (MDAS) was used to assess anxiety levels. The Modified Dental Anxiety Scale (MDAS) consisted of 5 questions ranging from 5 (no anxiety) to 25 (highest anxiety level). Every patient was asked to mark his or her perceived dental anxiety level on the line.
Evaluation of the relationship between patients' pretreatment anxiety levels and socio-demographic characteristics and dental treatment habits | Before Endodontic Treatment
  The patients were asked to fill in anxiety scales and sociodemographic/dental habits forms. State Anxiety Scale (STAI-S) was used to assess anxiety levels. The STAI-S scales consisted of two scales, each with 20 questions, with a total score between 20 and 80. Every patient was asked to mark his or her perceived dental anxiety level on the line.
Evaluation of the relationship between patients' pretreatment anxiety levels and socio-demographic characteristics and dental treatment habits | Before Endodontic Treatment
  The patients were asked to fill in anxiety scales and sociodemographic/dental habits forms. Trait Anxiety Scale (STAI-T) was used to assess anxiety levels. The STAI-T scales consisted of two scales, each with 20 questions, with a total score between 20 and 80. Every patient was asked to mark his or her perceived dental anxiety level on the line.
Evaluation of the relationship between patients' pretreatment anxiety levels and socio-demographic characteristics and dental treatment habits | Before Endodontic Treatment
  The patients were asked to fill in anxiety scales and sociodemographic/dental habits forms. The Visual Analogue Scale (VAS) was a scale consisting of a horizontal straight line 0-100 mm long with words describing the two extremes of the condition to be measured at both ends (i.e. zero - no anxiety, maximum - most severe anxiety). Every patient was asked to mark his or her perceived dental anxiety level on the line.

OTHER OUTCOMES:
Evaluation of patients satisfaction about information types | Immediately after treatment
  A feedback-satisfaction form containing 4 items about information types was applied to all patients after the endodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Dönmez Özkan, Study Director — Aydin Adnan Menderes University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Aydin Adnan Menderes University, Faculty of Dentistry, Department of Endodontics, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Najafpour E, Asl-Aminabadi N, Nuroloyuni S, Jamali Z, Shirazi S. Can galvanic skin conductance be used as an objective indicator of children's anxiety in the dental setting? J Clin Exp Dent. 2017 Mar 1;9(3):e377-e383. doi: 10.4317/jced.53419. eCollection 2017 Mar. PMID 28298978
- [Background] Caprara HJ, Eleazer PD, Barfield RD, Chavers S. Objective measurement of patient's dental anxiety by galvanic skin reaction. J Endod. 2003 Aug;29(8):493-6. doi: 10.1097/00004770-200308000-00001. PMID 12929693
- [Background] Kazancioglu HO, Tek M, Ezirganli S, Demirtas N. Does watching a video on third molar surgery increase patients' anxiety level? Oral Surg Oral Med Oral Pathol Oral Radiol. 2015 Mar;119(3):272-7. doi: 10.1016/j.oooo.2014.10.012. Epub 2014 Nov 8. PMID 25561389